CLINICAL TRIAL: NCT05968521
Title: Cardiac Rehabilitation for Young People: A Single-Blind Randomised Acceptability and Feasibility Study of an Integrated Physical and Mental Health Approach
Brief Title: Cardiac Rehabilitation for Young People
Acronym: CardioActive
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Greater Manchester Mental Health NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); University of Manchester (Other); University of York (Other)
Responsible Party: Principal Investigator, Lora Capobianco, Principal Investigator, Greater Manchester Mental Health NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: X638s
Record Dates: First submitted 2023-05-09; First posted 2023-08-01 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Congenital Heart Disease; Cardiomyopathies; Cardiac Arrythmias; Heart Failure; Cerebrovascular Event; Heart Valve Diseases
Keywords: Cardiac Rehabilitation; Metacognitive Therapy; Mental health; Feasibility; Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital; Cardiomyopathies; Heart Failure; Heart Valve Diseases; Psychological Well-Being | interventions — Cardiac Rehabilitation; Therapeutics

STUDY DESIGN:
Intervention Model Description: The study is a single blind parallel randomised feasibility trial comparing a CR programme against usual care with 100 CYP (50 per arm) aged 11-16 diagnosed with a heart condition.
Who Masked: Outcomes Assessor
Masking Description: Blinding of allocation will be maintained for the principal investigator's, statistician, and quantitative research assistant.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiac Rehabilitation (Intervention) (Experimental): Participants allocated to the intervention group will receive a cardiac rehabilitation (CR) programme which will involve education, exercise, and a psychological component.
  Interventions: Behavioral: Cardiac Rehabilitation (CR): Experimental
- Treatment as usual (Control) (Active Comparator): Participants allocated to the control group will receive treatment as usual.
  Interventions: Behavioral: Treatment as usual: Control

INTERVENTIONS:
Behavioral: Cardiac Rehabilitation (CR): Experimental — CR will consist of six sessions lasting 90 minutes of a structured exercise programme, educational and lifestyle modules, and a psychological component. Sessions include group discussions, experiential learning and homework tasks that participants are asked to complete between sessions. Participants in this treatment arm will also receive routine clinical outpatient management alongside CR.
  Arms: Cardiac Rehabilitation (Intervention)
Behavioral: Treatment as usual: Control — Treatment as usual will include routine clinical outpatient management.
  Arms: Treatment as usual (Control)

SUMMARY:
Heart problems are amongst the most common physical illnesses in children and young people (CYP). They can be present from birth or develop as CYP get older and are linked to increased physical and psychological difficulties overprotection from caregivers and healthcare providers and reduced quality of life.

While adults are offered exercise classes and lifestyle advice after a heart problem, CYP with heart problems are not. Improving health behaviours in people with heart problems is vital, improves quality of life and reduces additional illnesses (i.e obesity, diabetes).

Approximately 1 in 3 CYP with heart problems have anxiety and/or depression so it is also important to support their mental health. One way to do this is to develop and test the acceptability and feasibility of a trial of cardiac rehabilitation (CR) consisting of exercise with mental health support for CYP.

The aim is to develop and test the feasibility and acceptability of a trial of a cardiac rehabilitation programme for CYP.

ELIGIBILITY:
All participants meeting the following inclusion criteria and aged between 11-16 years old will be eligible:

Inclusion Criteria:

1. Fluent in English
2. Consent to participate
3. Diagnosed with at least one of the following:

   * Congenital heart disease (all subtypes)
   * Cardiomyopathy
   * Cardiac arrhythmia
   * Heart failure
   * Post-cerebrovascular event
   * Post-heart valve repair/replacement

Exclusion Criteria:

1. Significant risk or safeguarding concerns (i.e., suicidal ideation)
2. Head injury/organic impairment
3. Significant social and/or communication difficulties

Those with a formal diagnosis or under assessment for any above exclusion criteria will be excluded.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate (Feasibility Outcome) | Date of Baseline Assessment to end of follow-up (24 week follow up)
  Feasibility will be assessed using recruitment rate (i.e., number of patients consented and randomized, number of patients declined the study).
Retention Rate (Feasibility Outcome) | Date of Baseline Assessment to end of follow-up (24 week follow up)
  Feasibility will be assessed using retention rates (i.e., number of patients withdrawn from the study, lost to follow up)
Intervention Attendance (Feasibility Outcome) | Date of Baseline Assessment to end of follow-up (24 week follow up)
  Feasibility will be assessed using participant attendance at intervention (i.e., number of sessions attended at the intervention).
Acceptability of the Intervention | Date of Baseline Assessment to end of follow-up (24 week follow up)
  Acceptability of the intervention will be assessed in qualitative semi-structured interviews with children and young people, caregivers, and healthcare professionals, which will assess individuals views on the intervention, targets for improvement, and perceived acceptability of the components of the cardiac rehabilitation programme.

SECONDARY OUTCOMES:
Strength and Difficulties Questionnaire (SDQ) | Baseline, 12 weeks (end of treatment), and 24 weeks (follow-up)
  The SDQ measures psychological wellbeing across five subscales: emotion, hyperactivity, conduct, peer relations and pro-social behaviour. The SDQ can be completed by CYP and caregivers.
  Score for the subscales range from 0-10, with a total difficulties score (0-40) generated by summing together the scores from all subscales except the pro-social subscale. Higher scores on the pro-social scale reflect strengths whereas higher scores across other subscales reflect difficulties.
Paediatric Quality of Life (PedsQol) | Baseline, 12 weeks (end of treatment), and 24 weeks (follow-up)
  The PedsQol is a 23 item measures of health related quality of life, and includes four subscales: physical, emotional, social and school functioning. The questionnaire is commonly used in paediatric cardiology. The PedsQol will be completed by CYP.
  The items are scores from 0 (Never) to 4 (Almost always). Total scores range from 0-100, with higher scores indicating better quality of life.
Six minute walk test (6MWT) | Baseline, 12 weeks (end of treatment), and 24 weeks (follow-up)
  The 6MWT is used to assess aerobic capacity and endurance. Performance on the 6MWT has been predictive of morbidity and mortality whereby poorer performance is associated with increased mortality.
Incremental Shuttle Walk Test (ISWT) | Baseline, 12 weeks (end of treatment), and 24 weeks (follow-up)
  The ISWT is used to measure maximal exercise capacity. The ISWT is a 12-level test (1 min at each level), whereby participants walk up and down a 10, course with increasing accelearion of 0.17 m/s up to a maximum speed of 2.37 m/s. Walking speed is dicated by an audio signal. The test ends when the subject has a heart rate greater than 85% of their predicted maximum, is limited by dyspnoea or when the participant is unable to maintain the required speed and doe snot complete a shuttle for second consecutive time. The distance covered from the number of shuttles will be calculated.
Physical Activity Monitoring | Baseline, 12 weeks (end of treatment), and 24 weeks (follow-up)
  Participants will wear an accelerometer (Actigraph) for 5 days to monitor physical activity levels at each assessment.
Metacognition Questionnaire-Adolescent (MCQ-A) | Baseline, 12 weeks (end of treatment), and 24 weeks (follow-up)
  The MCQ-A assesses metacognitive beliefs (beliefs about thinking) across five subscales (uncontrollability of worry, need to control thoughts, cognitive self-consciousness, positive beliefs about worry, and cognitive confidence). The measure contains 30 items and is scored on a likert scale from 1 (do not agree) to 4 (agree very much). Total scores range from 30-120 and 6 to 30 for each subscale. Greater scores indicate greater maladaptive metacognitive beliefs.
  The measure and will be completed by CYP.
Child Health Utility-9D (CHU-9D) | Baseline, 12 weeks (end of treatment), and 24 weeks (follow-up)
  The CHU-9D measures quality of life using nine dimensions (worried, sad, pain, tired, annoyed, schoolwork/homework, sleep, daily routine, and ability to join in activities). Each item has 5 levels ranging from no problems to inability to do the item. Responses will be used to generate utility values in the health economic evaluation. The CHU-9D will be completed by CYP.
Health and Social Care Service-Use Questionnaire | Baseline, 12 weeks (end of treatment), and 24 weeks (follow-up)
  The questionnaire will include questions about whether the child has used any primary, secondary, or community-based health and social care and how often they used the service in the last 16 weeks (baseline study visit) or since the last assessment (follow-up study visits). The questionnaire will be developed from existing child relevant service use questionnaires held by the co-applicants and through discussion with the patient and public involvement representative, parent advisory group and clinical members of the study team. This will be completed by parents/primary caregivers. The responses given and the patient feedback will be used to further refine the health-resource use questionnaire ahead of the definitive study.
Demographics Questionnaire | Baseline, 12 weeks (end of treatment), and 24 weeks (follow-up)
  The demographics questionnaire will collect variables such as participants age, sex, weight, height, BMI, type of heart problem, comorbid mental and physical illnesses, ethnicity, medication, socioeconomic status, parental occupational status. This will be completed by the parents/primary caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Lora Capobianco, PhD, Principal Investigator — Greater Manchester Mental Health Foundation Trust; Adrian Wells, PhD, Principal Investigator — University of Manchester
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

REFERENCES:
- [Derived] Capobianco L, Hann M, McManus E, Peters S, Doherty PJ, Ciotti G, Murray J, Wells A. Cardiac rehabilitation for children and young people (CardioActive): protocol for a single-blind randomised feasibility and acceptability study of a centre-based cardiac rehabilitation programme versus usual care in 11-16 years with heart conditions. BMJ Open. 2024 Feb 24;14(2):e077958. doi: 10.1136/bmjopen-2023-077958. PMID 38401897